CLINICAL TRIAL: NCT06420843
Title: Microbiota, Metabolome and Nutrition: an 'Artificially Intelligent' Way to Personalized Nutrition
Acronym: PN-AI-21
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 3007
Record Dates: First submitted 2024-05-15; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: IBS - Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low FODMAP milk (Experimental): Patients will receive one week of low FODMAP diet supplemented with fermented milk followed by one week of low FODMAP diet supplemented with fermented beans.
  Interventions: Dietary Supplement: FOODMAP
- low FODMAP beans (Active Comparator): The second group will receive low FODMAP diet supplemented for one week with fermented beans followed by a second week of low FODMAP diet supplemented with fermented milk.
  Interventions: Dietary Supplement: FOODMAP

INTERVENTIONS:
Dietary Supplement: FOODMAP — Dietary restriction of fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAPs) have been recently investigated in the management of functional gut symptoms in IBS.

SUMMARY:
Intervention:

(Weeks 1-2, Visit 3-4) - Starting from the second week after the date of consent, patients with IBS will be randomized 1:1 into two groups. The first group (20 patients) will receive one week of a low FODMAP supplemented with fermented milk followed by one week of a low FODMAP content supplemented with fermented beans. The second group (20 patients) will receive a low FODMAP diet supplemented for one week with fermented beans followed by a second week of a diet with a low FODMAP diet supplemented with fermented milk. The microbiome of the patients will be evaluated after the first and second weeks along with data related to weight. After the second week, the metabolome and physical characteristics. The enrollment period will last for one year. The analysis of clinical data will be completed within one year after patient enrollment. Analysis of laboratory data will be performed in parallel.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a chronic intestinal condition whose high incidence and prevalence make it a major healthcare problem(3-7). IBS affects 7-15% of the general population(6, 7). It is twice as frequent in women(8) and is diagnosed more often in patients less than 50 years of age(9). It is characterized by recurrent episodes of functional gastrointestinal symptoms whose pathophysiological mechanisms are not completely clear(10). The most common symptoms include abdominal pain, bloating, constipation, and/or diarrhea(10). IBS negatively impacts quality of life and causes a substantial burden on healthcare resources(11, 12). Like the clinical phenotypes, the pathophysiological mechanisms underlying the syndrome are heterogeneous and not fully understood(13). However, there is evidence that IBS may result from a combination of gastrointestinal motility changes, visceral hypersensitivity, low-grade inflammation, altered microbiota, and food components(14-17). Due to the diversity of IBS symptoms and their considerable variability over time, a wide range of pharmacological treatments are employed which often only target the primary symptom; thus, when multiple symptoms are present, the treatments administered are often inadequate. This has led to the investigation of use of dietary therapies as a treatment option.

Dietary restriction of fermentable oligosaccharides, disaccharides, monosaccharides and polyols (FODMAPs) have been recently investigated in the management of functional gut symptoms in IBS. An increasing number of uncontrolled and controlled trials have examined the clinical effectiveness of a low FODMAP diet in patients with IBS using either dietary advice or feeding protocols. Uncontrolled and unblinded controlled trials suggest symptom response rates in patients with IBS are as high as 85%(18). Similarly, a beneficial impact on symptoms has been reported in blinded randomized controlled trials(19-22). A potential shortcoming of the low FODMAP diet and of any diet that involves multiple food exclusion, is the risk of nutritional inadequacy, and this is especially pertinent if the excluded foods are nutrient-rich. The low FODMAP diet requires substitution of selected food items across a number of food groups and, therefore, there is the potential for inadequate intake of nutrients, particularly carbohydrate, fiber, iron, B vitamins, and calcium. Another potential safety concern associated with implementation of the diet relates to the impact on the gastrointestinal microbiota, which has been implicated in the pathogenesis of IBS(23) and has been associated with clinical features of IBS including abdominal pain, anxiety, and depression(24, 25). Hence, we propose to evaluate the microbiome and metabolome in IBS patients to create datasets of integrated data through AI tools. Furthermore, we aim to determine the effects of a low FOODMAP diet based on fermented products on the microbiome and metabolome in IBS patients. These evaluations will allow to assess patient's nutrient deficiency and the general quality of life pre and post intervention among groups and to develop a personalized treatment that will increase the quality of life in IBS patients.

The low FODMAPs diet is associated with limitations particularly due to the elimination of several food items which can cause worsening of the side effects due to significant alteration of the intestinal microbiota composition and an overall reduction of the nutritional status. Although, probiotics seem to have beneficial effects on improving this side effect, their way of function is still relatively unknown. Much remains to be answered as to which strains is/are most effective across the broad spectrum of IBS patients and whether single or combination of strains work best. This leads to the question of whether individual differences among IBS patients in terms of microbiome diversity could affect the efficacy of probiotics therapy. Therefore, with our approach we propose a reshaping of the host-microbiota interactions through personalized nutrition which could be a new therapeutic avenue for both disease control and prevention. Specifically, we believe that a diet supplemented with previously fermented food items will be beneficial for the patient's condition. This fermentation will be controlled and performed with Lactobacillus paracasei strain CNCM I-5220. Through the longitudinal study we will be able to evaluate their grade of the disorder at baseline (one week of low FODMAP diet), and the effect of the fermented food items on their microbiota and metabolome after one and two weeks. Furthermore, by adopting new efficacious treatment options, it might be possible to decrease the high recurrence rate of IBS patients to the public health system, improving patient's quality of life and decreasing the costs for the National Sanitary System (SSN).

The primary objective will be to assess the enterotypes of IBS patient at baseline and to analyze how supplementation of fermented food modifies the microbiome and metabolome in IBS patients following a low FODMAP diet.

As secondary objective, we will compare the efficacy and safety of two different nutritional approaches on IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sex and any race
* Age ≥18 and ≤70.
* IBS confirmed by Rome IV diagnostic criteria
* Willing to adhere to the proposed diet
* Provision of written informed consent
* Commitment of availability throughout the study period

Exclusion Criteria:

* Patient age <18 and > 70
* Diabetes (Type 1 or 2)
* Subjects who have used probiotic, antibiotic, lactic ferment or pump inhibitors within 15 days prior to screening.
* Pregnant or planning to become pregnant or is lactating.
* History of HIV or hepatitis B or C
* Participation in investigational study within past 30 days
* Unstable cardiovascular or pulmonary disease, with change in treatment in last 30 days due to worsening disease condition
* Any concomitant disease requiring specialized nutrition (e.g. renal failure, celiac disease, cerebrovascular disease of the central nervous system, major surgical cavity)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-12-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome | 1 week
  The primary endpoint will be the change in the phenotype of microbiome and metabolome in the two-study group at the end of the assumption of fermented food. Stool samples will be thoroughly analyzed for microbiome (amplified for 16S rDNA sequencing and/or shotgun) and metabolome composition (untargeted). IBS-related symptoms will also be evaluated at the end of one week of low FODMAP diet consumption.

SECONDARY OUTCOMES:
Microbiome after baseline | 2 weeks
  to assess and compare the changes in the microbiome and metabolome phenotype at baseline and 1 week after the low FODMAP diet assumption, and after 1 week of addition of fermented food.Patients' microbiome will be assessed after the first and second week by collecting a fecal sample together with data regarding the weight. Metabolome and IBS-related symptoms will be evaluated in a longitudinal study after the second week as previously mentioned.
GSRS score | 1 week
  to assess and compare any change in the GSRS score at baseline, after 1 week of low FODMAP diet assumption and at the end of the study in the two study groups.
  GSRS is a symptom assessment tool that measures the baseline severity and frequency of these symptoms, as well as the response to treatment(1).

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Gastroenterology Department, Humanitas Research Hospital, Rozzano, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Svedlund J, Sjodin I, Dotevall G. GSRS--a clinical rating scale for gastrointestinal symptoms in patients with irritable bowel syndrome and peptic ulcer disease. Dig Dis Sci. 1988 Feb;33(2):129-34. doi: 10.1007/BF01535722. PMID 3123181
- [Background] Gibson PR, Shepherd SJ. Evidence-based dietary management of functional gastrointestinal symptoms: The FODMAP approach. J Gastroenterol Hepatol. 2010 Feb;25(2):252-8. doi: 10.1111/j.1440-1746.2009.06149.x. PMID 20136989
- [Background] Altobelli E, Lattanzi A, Paduano R, Varassi G, di Orio F. Colorectal cancer prevention in Europe: burden of disease and status of screening programs. Prev Med. 2014 May;62:132-41. doi: 10.1016/j.ypmed.2014.02.010. Epub 2014 Feb 14. PMID 24530610
- [Background] Altobelli E, D'Aloisio F, Angeletti PM. Colorectal cancer screening in countries of European Council outside of the EU-28. World J Gastroenterol. 2016 May 28;22(20):4946-57. doi: 10.3748/wjg.v22.i20.4946. PMID 27239121
- [Background] Burisch J, Jess T, Martinato M, Lakatos PL; ECCO -EpiCom. The burden of inflammatory bowel disease in Europe. J Crohns Colitis. 2013 May;7(4):322-37. doi: 10.1016/j.crohns.2013.01.010. Epub 2013 Feb 8. PMID 23395397
- [Background] American College of Gastroenterology Task Force on Irritable Bowel Syndrome; Brandt LJ, Chey WD, Foxx-Orenstein AE, Schiller LR, Schoenfeld PS, Spiegel BM, Talley NJ, Quigley EM. An evidence-based position statement on the management of irritable bowel syndrome. Am J Gastroenterol. 2009 Jan;104 Suppl 1:S1-35. doi: 10.1038/ajg.2008.122. No abstract available. PMID 19521341
- [Background] Andrews EB, Eaton SC, Hollis KA, Hopkins JS, Ameen V, Hamm LR, Cook SF, Tennis P, Mangel AW. Prevalence and demographics of irritable bowel syndrome: results from a large web-based survey. Aliment Pharmacol Ther. 2005 Nov 15;22(10):935-42. doi: 10.1111/j.1365-2036.2005.02671.x. PMID 16268967
- [Background] Muller-Lissner SA, Bollani S, Brummer RJ, Coremans G, Dapoigny M, Marshall JK, Muris JW, Oberndorff-Klein Wolthuis A, Pace F, Rodrigo L, Stockbrugger R, Vatn MH. Epidemiological aspects of irritable bowel syndrome in Europe and North America. Digestion. 2001;64(3):200-4. doi: 10.1159/000048862. PMID 11786669
- [Background] El-Salhy M, Gundersen D, Gilja OH, Hatlebakk JG, Hausken T. Is irritable bowel syndrome an organic disorder? World J Gastroenterol. 2014 Jan 14;20(2):384-400. doi: 10.3748/wjg.v20.i2.384. PMID 24574708
- [Background] Horwitz BJ, Fisher RS. The irritable bowel syndrome. N Engl J Med. 2001 Jun 14;344(24):1846-50. doi: 10.1056/NEJM200106143442407. No abstract available. PMID 11407347
- [Background] Chang L. Review article: epidemiology and quality of life in functional gastrointestinal disorders. Aliment Pharmacol Ther. 2004 Nov;20 Suppl 7:31-9. doi: 10.1111/j.1365-2036.2004.02183.x. PMID 15521853
- [Background] Maxion-Bergemann S, Thielecke F, Abel F, Bergemann R. Costs of irritable bowel syndrome in the UK and US. Pharmacoeconomics. 2006;24(1):21-37. doi: 10.2165/00019053-200624010-00002. PMID 16445300
- [Background] Chey WD, Kurlander J, Eswaran S. Irritable bowel syndrome: a clinical review. JAMA. 2015 Mar 3;313(9):949-58. doi: 10.1001/jama.2015.0954. PMID 25734736
- [Background] Anastasi JK, Capili B, Chang M. Managing irritable bowel syndrome. Am J Nurs. 2013 Jul;113(7):42-52; quiz 54, 53. doi: 10.1097/01.NAJ.0000431911.65473.35. PMID 23764698
- [Background] Mayer EA. Clinical practice. Irritable bowel syndrome. N Engl J Med. 2008 Apr 17;358(16):1692-9. doi: 10.1056/NEJMcp0801447. PMID 18420501
- [Background] Mayer EA, Labus JS, Tillisch K, Cole SW, Baldi P. Towards a systems view of IBS. Nat Rev Gastroenterol Hepatol. 2015 Oct;12(10):592-605. doi: 10.1038/nrgastro.2015.121. Epub 2015 Aug 25. PMID 26303675
- [Background] Rajilic-Stojanovic M, Jonkers DM, Salonen A, Hanevik K, Raes J, Jalanka J, de Vos WM, Manichanh C, Golic N, Enck P, Philippou E, Iraqi FA, Clarke G, Spiller RC, Penders J. Intestinal microbiota and diet in IBS: causes, consequences, or epiphenomena? Am J Gastroenterol. 2015 Feb;110(2):278-87. doi: 10.1038/ajg.2014.427. Epub 2015 Jan 27. PMID 25623659
- [Background] Staudacher HM, Irving PM, Lomer MC, Whelan K. Mechanisms and efficacy of dietary FODMAP restriction in IBS. Nat Rev Gastroenterol Hepatol. 2014 Apr;11(4):256-66. doi: 10.1038/nrgastro.2013.259. Epub 2014 Jan 21. PMID 24445613
- [Background] Staudacher HM, Lomer MC, Anderson JL, Barrett JS, Muir JG, Irving PM, Whelan K. Fermentable carbohydrate restriction reduces luminal bifidobacteria and gastrointestinal symptoms in patients with irritable bowel syndrome. J Nutr. 2012 Aug;142(8):1510-8. doi: 10.3945/jn.112.159285. Epub 2012 Jun 27. PMID 22739368
- [Background] Halmos EP, Power VA, Shepherd SJ, Gibson PR, Muir JG. A diet low in FODMAPs reduces symptoms of irritable bowel syndrome. Gastroenterology. 2014 Jan;146(1):67-75.e5. doi: 10.1053/j.gastro.2013.09.046. Epub 2013 Sep 25. PMID 24076059
- [Background] Bohn L, Storsrud S, Liljebo T, Collin L, Lindfors P, Tornblom H, Simren M. Diet low in FODMAPs reduces symptoms of irritable bowel syndrome as well as traditional dietary advice: a randomized controlled trial. Gastroenterology. 2015 Nov;149(6):1399-1407.e2. doi: 10.1053/j.gastro.2015.07.054. Epub 2015 Aug 5. PMID 26255043
- [Background] Eswaran SL, Chey WD, Han-Markey T, Ball S, Jackson K. A Randomized Controlled Trial Comparing the Low FODMAP Diet vs. Modified NICE Guidelines in US Adults with IBS-D. Am J Gastroenterol. 2016 Dec;111(12):1824-1832. doi: 10.1038/ajg.2016.434. Epub 2016 Oct 11. PMID 27725652
- [Background] Simren M, Barbara G, Flint HJ, Spiegel BM, Spiller RC, Vanner S, Verdu EF, Whorwell PJ, Zoetendal EG; Rome Foundation Committee. Intestinal microbiota in functional bowel disorders: a Rome foundation report. Gut. 2013 Jan;62(1):159-76. doi: 10.1136/gutjnl-2012-302167. Epub 2012 Jun 22. PMID 22730468
- [Background] Sundin J, Rangel I, Fuentes S, Heikamp-de Jong I, Hultgren-Hornquist E, de Vos WM, Brummer RJ. Altered faecal and mucosal microbial composition in post-infectious irritable bowel syndrome patients correlates with mucosal lymphocyte phenotypes and psychological distress. Aliment Pharmacol Ther. 2015 Feb;41(4):342-51. doi: 10.1111/apt.13055. Epub 2014 Dec 18. PMID 25521822
- [Background] Parkes GC, Rayment NB, Hudspith BN, Petrovska L, Lomer MC, Brostoff J, Whelan K, Sanderson JD. Distinct microbial populations exist in the mucosa-associated microbiota of sub-groups of irritable bowel syndrome. Neurogastroenterol Motil. 2012 Jan;24(1):31-9. doi: 10.1111/j.1365-2982.2011.01803.x. Epub 2011 Nov 9. PMID 22070725
- [Background] Pasolli E, Truong DT, Malik F, Waldron L, Segata N. Machine Learning Meta-analysis of Large Metagenomic Datasets: Tools and Biological Insights. PLoS Comput Biol. 2016 Jul 11;12(7):e1004977. doi: 10.1371/journal.pcbi.1004977. eCollection 2016 Jul. PMID 27400279
- [Background] Troisi J, Sarno L, Landolfi A, Scala G, Martinelli P, Venturella R, Di Cello A, Zullo F, Guida M. Metabolomic Signature of Endometrial Cancer. J Proteome Res. 2018 Feb 2;17(2):804-812. doi: 10.1021/acs.jproteome.7b00503. Epub 2018 Jan 2. PMID 29235868
- [Background] Bar-Joseph Z, Gifford DK, Jaakkola TS. Fast optimal leaf ordering for hierarchical clustering. Bioinformatics. 2001;17 Suppl 1:S22-9. doi: 10.1093/bioinformatics/17.suppl_1.s22. PMID 11472989